CLINICAL TRIAL: NCT06511531
Title: Clinical Features and Possible Mechanisms in Patients With Sarcopenia in Parkinson's Disease
Brief Title: Exploring Sarcopenia in Parkinson's Disease Patients by Combining Serum Biomarker Levels
Status: Not yet recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Lixia Qin, Principal Investigator, Central South University
Other Study IDs: Xiangya_PD and Sarcopenia
Record Dates: First submitted 2024-06-22; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's Disease (PD) and sarcopenia are prevalent age-related syndromes, often occurring simultaneously within individuals. Sarcopenia is notably common among PD patients, with severe cases affecting approximately one in every five individuals with PD. Moreover, sarcopenia is closely linked to the accelerated progression of PD, diminished quality of life, heightened mortality risk, and increased susceptibility to falls and fractures. Therefore, early detection of sarcopenia assumes particular significance as it offers an opportunity for interventions aimed at mitigating or delaying muscle degeneration, potentially influencing PD outcomes. This review will delve into the relationship between sarcopenia and PD, methods for screening and testing sarcopenia, and potential avenues for further research and the development of strategies for risk reduction and treatment

DETAILED DESCRIPTION:
The onset of sarcopenia in PD may be intricately linked to both motor and non-motor symptoms. In terms of motor symptoms, sarcopenia exacerbates muscle weakness, impairs balance and gait, and may worsen symptoms like rigidity and bradykinesia in PD. Numerous studies have shown that sarcopenia is strongly associated with disease duration, Hoehn-Yahr staging, and Unified PD Rating Scale-III(UPDRSIII) scores. Regarding non-motor symptoms, sarcopenia contributes to increased fatigue due to muscle weakness, disrupts sleep patterns, exacerbates psychological distress including depression and anxiety, and may impact cognitive function. In addition, some studies supported that the incidence of falls, disability and death in PD with Sarcopenia were higher than those in PD without sarcopenia.

Nevertheless, other studies have reported controversial results. Some researchers believed that sarcopenia had no correlations with disease duration, HY, UPDRS-I/III, cognition and depression. However, most of the current studies are small cross-sectional studies that are not very convincing about the relationship between diseases. Thus, further studies with long-term follow up and large sample sizes are required to determine the causal direction of these relationships.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as either ''definite'' or ''probable'' PD based on Chinese diagnostic criteria of Parkinson's disease (2016 version)

Exclusion Criteria:

Parkinson's syndrome or Parkinsonian superimposed syndrome due to encephalitis, cerebrovascular disease, poisoning, trauma, drugs or other factors

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 30 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
the SARC-F | 12 months
  The SARC-F is a simple screening tool for sarcopenia, consisting of five questions on strength, assistance in walking, rising from a chair, climbing stairs, and falls. Each question is scored from 0 to 2, with a total score of 4 or more indicating a risk of sarcopenia.

SECONDARY OUTCOMES:
Low Muscle Mass | 12 months
  The Skeletal Muscle Mass Index (SMI) is a measure used to assess muscle mass relative to a person's height. It is calculated by dividing the total skeletal muscle mass (usually obtained through techniques like DXA or BIA) by the square of the individual's height (in meters)
Low Muscle Strength | 12 months
  Commonly assessed using grip strength tests
Poor Physical Performance | 12 months
  Evaluated through tests like gait speed, the Short Physical Performance Battery (SPPB), or the Timed Up and Go (TUG) test.